CLINICAL TRIAL: NCT05873764
Title: [14C] -RV521.HCl - A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion Following a Single Oral Dose in Healthy Male Subjects
Brief Title: A Study to Learn About Effect of Sisunatovir in Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REVC008; C5241008 (Other: Alias Study Number)
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 200 mg RV521/78 µCi [ 14C]-RV521 (Experimental): 200 mg RV521/78 µCi [ 14C]-RV521
  Interventions: Drug: 200 mg RV521/78 µCi [ 14C]-RV521.

INTERVENTIONS:
Drug: 200 mg RV521/78 µCi [ 14C]-RV521. — 200 mg RV521/78 µCi [ 14C]-RV521

SUMMARY:
The purpose of this clinical trial is to learn about the safety, effects, and tolerability of the study medicine (sisunatovir).

This study is looking for healthy adult participants who meet the following criteria:

1. Males age 18 to 55 years
2. All fertile participants must agree to the use of highly effective contraception
3. Body mass index (BMI) of 18 to 32.0 kg/m2; body weight of 55.0 to 100.0 kg.
4. Participants who are overtly healthy as determined by medical evaluation. This includes medical history, physical examination, blood pressure, pulse rate, standard 12-lead ECG (electrocardiogram), and laboratory tests.

This study will enroll up to 10 participants. All study participants will receive 1 dose of sisunatovir by mouth. The study duration is expected to be about 9 weeks. This includes a 28-day screening period, 16-day inpatient stay, and 2 overnight follow-up visits, if needed.

ELIGIBILITY:
Inclusion Criteria (key):

* Males
* Age 18- 55 years
* Body mass index (BMI) 18.0 kg/m2 to 32.0 kg/m2
* Body weight 55.0 kg to 100.0 kg
* Considered to be in good health
* Nonsmoker
* Content of 14C in urine, whole blood, and/or plasma samples does not exceed the general environmental background level of 14C

Exclusion Criteria (key):

* Clinically significant abnormal medical history or any abnormal finding on physical examination, vital signs, ECG, laboratory tests
* History of cancer that has not been in full remission for >5 years
* Acute illness within 14 days prior to Day 1
* History of significant drug allergies
* History or presence of alcohol or drug abuse
* Recent history of incomplete bladder emptying with voiding or awakening more than once at night to void
* Usual habit of <1 or >3 bowel movements per day
* Exposure to radiation for therapeutic, diagnostic, or occupational reasons within the 12 months prior to Day 1.
* Participation in another clinical study in which a [14C]-labeled drug was administered within 1 year prior to Check-in
* Administration of another investigational medication within 60 days (or 5 half-lives, whichever is longer) prior to Day 1
* Participation in an investigational-device study within 60 days prior to Day 1
* Any ECG abnormality considered to be clinically significant by the Investigator
* QTcF interval >450 msec and QRS interval >120 msec
* Family history of long QT syndrome or of unexplained sudden death in a first-degree relative under 50 years of age
* Documented congenital or acquired long QT syndrome
* Presence of clinically significant hypertension
* Presence of clinically significant hypotension
* Loss or donation of more than 500 mL blood within 60 days prior to the Screening
* Excessive consumption of alcohol
* Use of any live vaccinations within 30 days
* Use/consumption of food or drugs known to be moderate or strong cytochrome P450 3A4 (CYP3A4) inducers or potent CYP3A4 inhibitors within 14 days or 5 half-lives, whichever is longer, prior to RV521 administration

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Tmax (Time of maximum observed concentration) | Day 1 (time 0) to Day 29
  PK parameters of total radioactivity and RV521 following a single oral administration of [ 14C]-RV521 to healthy male subjects
Cmax (Maximum observed concentration) | Day 1 (time 0) to Day 29
  PK parameters of total radioactivity and RV521 following a single oral administration of [ 14C]-RV521 to healthy male subjects
AUC0-inf (Area under the concentration-time curve (AUC) extrapolated to infinity) | Day 1 (time 0) to Day 29
  PK parameters of total radioactivity and RV521 following a single oral administration of [ 14C]-RV521 to healthy male subjects
AUC0-last (AUC from the time of dosing to the time of the last measurable concentration) | Day 1 (time 0) to Day 29
  PK parameters of total radioactivity and RV521 following a single oral administration of [ 14C]-RV521 to healthy male subjects
lambdaz (Rate constant associated with the terminal elimination phase) | Day 1 (time 0) to Day 29
  PK parameters of total radioactivity and RV521 following a single oral administration of [ 14C]-RV521 to healthy male subjects
t1/2 (half-life of the terminal elimination phase) | Day 1 (time 0) to Day 29
  PK parameters of total radioactivity and RV521 following a single oral administration of [ 14C]-RV521 to healthy male subjects
CL/F (Apparent clearance of the drug from plasma after oral administration) | Day 1 (time 0) to Day 29
  PK parameters of total radioactivity and RV521 following a single oral administration of [ 14C]-RV521 to healthy male subjects
Vz/F (Volume of distribution associated with the terminal phase) | Day 1 (time 0) to Day 29
  PK parameters of total radioactivity and RV521 following a single oral administration of [ 14C]-RV521 to healthy male subjects
CLR (renal clearance) | Day 1 (time 0) to Day 29
  PK parameters of total radioactivity and RV521 following a single oral administration of [ 14C]-RV521 to healthy male subjects
Fe (fraction of administered drug excreted into urine) | Day 1 (time 0) to Day 29
  PK parameters of total radioactivity and RV521 following a single oral administration of [ 14C]-RV521 to healthy male subjects
Ae0-t (cumulative amount of 14C excreted into urine from time 0 to the last sampling interval) | Day 1 (time 0) to Day 29
  PK parameters of total radioactivity and RV521 following a single oral administration of [ 14C]-RV521 to healthy male subjects
Ae0-t (Cumulative amount of 14C excreted into urine and feces from time 0 to the last sampling interval (in units of mass-equivalents/g)) | Day 1 (time 0) to Day 29
  Mass balance parameters in urinary and fecal excretion of radioactivity
Aet (Amount of 14C excreted into urine and feces per sampling interval (in units of mass-equivalents/g)) | Day 1 (time 0) to Day 29
  Mass balance parameters in urinary and fecal excretion of radioactivity
Fet (Fraction of 14C excreted into urine and feces per sampling interval (in units of %)) | Day 1 (time 0) to Day 29
  Mass balance parameters in urinary and fecal excretion of radioactivity
Fe0-t (Cumulative fraction of 14C excreted into urine or feces from time 0) | Day 1 (time 0) to Day 29
  Mass balance parameters in urinary and fecal excretion of radioactivity
14C associated with % of AUC of the total in plasma | Day 1 (time 0) to Day 29
  Metabolite Profiling and Identification
14C associated with % of administered dose of the total in urine and feces | Day 1 (time 0) to Day 29
  Metabolite Profiling and Identification

SECONDARY OUTCOMES:
Spontaneously reported adverse events (AEs) during the Treatment Period | Day -1 to Day 29
  safety and tolerability of a single oral dose of RV521 in healthy male subjects
Spontaneously reported serious AEs (SAEs) during the Treatment Period | Day -1 to Day 29
  Safety and tolerability of a single oral dose of RV521 in healthy male subjects
Use of concomitant medications | Day -1 to Day 29
  Safety and tolerability of a single oral dose of RV521 in healthy male subjects
Unscheduled assessments as needed for management of AEs | Day -1 to Day 29
  Safety and tolerability of a single oral dose of RV521 in healthy male subjects
Clinically significant changes from baseline of any of the following: Vital Signs (blood pressure, heart rate [HR], respiratory rate [RR], and oral temperature) | Day -1 to Day 29
  Safety and tolerability of a single oral dose of RV521 in healthy male subjects
Clinically significant changes from baseline of any of the following: 12-lead electrocardiogram (ECD) assessments | Day -1 to Day 29
  Safety and tolerability of a single oral dose of RV521 in healthy male subjects
Clinically significant changes from baseline of any of the following: Physical examinations | Day -1 to Day 29
  Safety and tolerability of a single oral dose of RV521 in healthy male subjects
Blood/Plasma AUC Ratio | Day 1 (time 0 to Day 29)
  AUC0-inf of total 14C in whole blood divided by the AUC0-inf of total 14C in plasma
Amount of 14C excreted into nostrils per sampling interval (in units of mass-equivalents/g) | Day 1 (time 0) to Day 29
  Metabolite Profiling and Identification
Cumulative amount of 14C excreted into nostrils, urine, and feces from time 0 to the last sampling interval (in units of mass-equivalents/g) | Day 1 (time 0 to Day 29)
  Metabolite Profiling and Identification
Evaluation of total radioactivity in nasal samples following a single oral administration of [ 14C]-RV521 to healthy male subjects | Day 1 (time 0) to Day 29
  PK parameters of total radioactivity and RV521 following a single oral administration of [ 14C]-RV521 to healthy male subjects
Structural identification of major metabolites | Day 1 (time 0) to Day 29
  Identification of each metabolite that accounts for ≥10% of circulating radiolabel

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pharmaron Clinical Pharmacology Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=REVC008